CLINICAL TRIAL: NCT02546947
Title: Monitoring in Intensive Care Unit of Neuromuscular Blocking Agents (NMBA) Used for Acute Respiratory Distress Syndrome (ARDS) After Cardiothoracic Surgery
Brief Title: Monitoring in Intensive Care Unit of Neuromuscular Blocking Agents Used for Acute Respiratory Distress Syndrome After Cardiothoracic Surgery
Acronym: CURAREA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Chirurgical Marie Lannelongue (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2013-A00067-38
Record Dates: First submitted 2015-08-27; First posted 2015-09-11 (Estimated); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Acute Respiratory Distress Syndrome
Keywords: Respiratory Distress Syndrome, Adult; Neuromuscular Blocking Agents; Atracurium; Mechanical ventilation; ARDS; partial pressure of oxygen(PaO2) /inspired oxygen (FiO2) < 200; Positive End Expiratory Pressure (PEEP) > 5 since less than 48 hrs
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Appropriate clinical group (No Intervention): group of patients with clinical dose adjustment
- TOF adapted group (Active Comparator): group with an objective of less than 2 responses to TOF stimulation monitored
  Interventions: Other: Train of four monitoring

INTERVENTIONS:
Other: Train of four monitoring — with an end point of one or two response at orbicularis oculi to TOF stimulation
  Arms: TOF adapted group

SUMMARY:
Mortality in Acute Respiratory Distress Syndrome (ARDS) is high (40 to 60 %). Protective mechanical ventilation is the cornerstone of the ARDS therapeutic strategies. Recently, a prospective multicenter study demonstrates that short-term infusion of neuromuscular blocking agents (NMBA) reduces hospital mortality. However, the mechanisms through which NMBAs could improve survival remain speculative and the dose of NMBA needed to observe a beneficial effect is still debated. In hypoxemic ventilated patients, continuous cisatracurium infusion with an objective of no response at orbicularis oculi to train-of-four (TOF) stimulation and an objective of two responses had similar effects on respiratory parameters. In their study, Papazian and colleagues used cisatracurium with an initial standard dose of 15 mg followed by a continuous infusion of 37.5mg/h, based on previous results of studies with patients monitored for paralysis. Atracurium and its stereoisomer cisatracurium are non-depolarizing neuromuscular blocking drugs, both used in anaesthesia and intensive care units.

The aim of this study was to compare in ARDS patients a dose adjustment of continuous-atracurium intravenous infusion with an end point of one or two response at orbicularis oculi to TOF stimulation, and a dose adjustment to achieve clinical goals of protective ventilation without monitoring of TOF stimulation.

ELIGIBILITY:
Inclusion Criteria:

* ARDS with a PaO2 / FiO2 < 200 with a PEEP > 5 since less than 48 hrs
* Informed consent

Exclusion Criteria:

* NMBA allergy
* Continuous administration of NMBA for ARDS prior inclusion
* Age < 18 yrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
cumulative total dose of atracurium (mg per kg per hour, administered from the initial phase of ARDS until disruption ≥48 hours) | 2 years
  was the primary outcome, calculated by the following formula:(Initial bolus dose +(standard bolus dose x number of repetition doses)+cumulative continuous infusion dose (mg/h x number of hours))/ weight (kg) x duration of administration (hour).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Chirurgical Marie Lannelongue, Le Plessis-Robinson, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rezaiguia-Delclaux S, Laverdure F, Genty T, Imbert A, Pilorge C, Amaru P, Sarfati C, Stephan F. Neuromuscular Blockade Monitoring in Acute Respiratory Distress Syndrome: Randomized Controlled Trial of Clinical Assessment Alone or With Peripheral Nerve Stimulation. Anesth Analg. 2021 Apr 1;132(4):1051-1059. doi: 10.1213/ANE.0000000000005174. PMID 33002927